CLINICAL TRIAL: NCT03098446
Title: The Effect of Sitting and Moderate Exercise on Plasma Triglyceride Elevation After a Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Edward F. Coyle, Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2016-12-0022
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Atherosclerosis; Metabolic Syndrome
MeSH Terms: conditions — Atherosclerosis; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either the sitting plus exercise or the sitting without exercise group and then, after a one week washout period, complete the other task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged sitting with exercise (Experimental): Subjects will be asked to undergo prolonged sitting (~14-hours/day) for 4 days. On the evening of day 4, they will be asked to run at 65% of VO2max for 1-hour.
  Interventions: Behavioral: Prolonged sitting with exercise
- Prolonged sitting without exercise (Experimental): Subjects will be asked to undergo prolonged sitting (~14-hours/day) for 4 days. Subjects will not be asked to complete the acute bout of exercise to serve as a control.
  Interventions: Behavioral: Prolonged sitting without exercise

INTERVENTIONS:
Behavioral: Prolonged sitting with exercise — Subjects will have a 2-day control period during which step count and diet will be controlled for and recreated for the other trial. Following this 2-day period, they will undergo the prolonged sitting trial with the acute bout of exercise on day 4. Day 5 will consist of the lipid tolerance test to determine the ability of the body to clear triglycerides.
  Arms: Prolonged sitting with exercise
Behavioral: Prolonged sitting without exercise — Subjects will have a 2-day control period during which step count and diet will be controlled for and recreated for the other trial. Following this 2-day period, they will undergo the prolonged sitting trial, but will not be asked to complete an acute bout of exercise on day 4. Day 5 will consist of the lipid tolerance test to determine the ability of the body to clear triglycerides.
  Arms: Prolonged sitting without exercise

SUMMARY:
The purpose of this study is to investigate the effect of 4 days of sitting and moderate exercise on plasma triglyceride elevation after a meal.

DETAILED DESCRIPTION:
Subjects will undergo three weeks (two intervention, one washout) of testing during which they will participate in two conditions: 1) prolonged sitting (~14-hours/day) with a 1-hour bout of acute exercise at 65% of pre-intervention VO2max and 2) prolonged sitting (~14-hours/day) without an acute bout of exercise. During each intervention week, subjects will have 2 days of dietary and activity control, followed by 4 days during which prolonged sitting will occur. On the evening of the 4th day, subjects in the exercise group will perform the acute bout of exercise. On day 5, all subjects will undergo a lipid tolerance test to determine the body's ability to clear triglycerides from the blood as well as insulin/glucose response and substrate oxidation. Blood samples will be assayed for the previously mentioned substances and postprandial gas collection will be analyzed via indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* cardiovascular problems (e.g. pre-existing heart issues, coronary artery disease, hypertension, etc.)
* respiratory problems
* musculoskeletal problems that prevent prolonged sitting or exercise
* obesity
* susceptibility to fainting

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-08 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Plasma Triglycerides | 6-hours
  Areas under the curve for triglyceride concentration will be calculated for hourly samples from a 6-hour lipid tolerance test

SECONDARY OUTCOMES:
Plasma Insulin | 6-hours
  Areas under the curve for insulin concentration will be calculated for hourly samples from a 6-hour lipid tolerance test
Plasma Glucose | 6-hours
  Areas under the curve for glucose concentration will be calculated for hourly samples from a 6-hour lipid tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin Human Performance Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No